CLINICAL TRIAL: NCT00796432
Title: Open-label Positron Emission Tomography (PET) Study of Central D2-receptor Occupancy in Healthy Subjects Following a Single Oral Dose of OROS Paliperidone
Brief Title: A Study of Dopamine Type 2 (D2) Receptor Occupancy Following a Single Oral Dose of OROS Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004267
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; mood disorders; antipsychotic drugs; dopamine; receptor occupancy; OROS paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: OROS paliperidone

SUMMARY:
The purposes of this study are to estimate the relationship of D2-receptor occupancy to plasma concentration and to assess the safety of OROS paliperidone.

DETAILED DESCRIPTION:
This is a single-center, single-dose, open-label, Phase-1 Positron Emission Tomography (PET) study in 4 healthy volunteers, 2 men and 2 women. After screening, healthy eligible volunteers will be hospitalized in the study unit from study Day 2 to Day 4. On Day 1 (the day before hospitalization), volunteers will enter the study unit from 5:00 p.m. to 8:00 p.m. for baseline prolactin blood sampling and sedation assessment. Each volunteer will have a control magnetic resonance imaging (at screening) and 3 PET measurements using the radioligand [11]C raclopride to measure central D2 receptor occupancy in the putamen. Blood samples to measure plasma concentrations of paliperidone will be collect immediately before and at scheduled time points after dose administration on Day 2, and immediately before, halfway through, and immediately after the PET-2 and PET-3 measurements. Serum prolactin levels will be measured immediately before and at several scheduled time points after dose administration, and immediately before and after each PET measurement. At scheduled time points, supine and standing blood pressures, pulse, sensorium changes, temperature, and degree of sedation will be recorded, volunteers will be questioned about adverse events, and they will be evaluated for extrapyramidal symptoms (EPS). Adverse events will be recorded and followed throughout the study. The rationale for the study design is based on previous PET studies with risperidone, which indicated that PET measurement of D2 receptor occupancy after a single dose of medication is useful in predicting an effective clinical dose range. Single oral dose (6 mg) of OROS paliperidone

ELIGIBILITY:
Inclusion Criteria:

* Within 20% of ideal body weight
* If a woman, must be surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, male partner sterilization) before entry and throughout the study
* and must have a negative serum beta HCG test at screening
* Healthy on the basis of a pre-study physical examination, medical history, anamnesis, electrocardiogram, magnetic resonance imaging of the brain, and the results of blood biochemistry and hematology tests and a urinalysis carried out less than 2 weeks before the first dose. If the results of the biochemistry or hematology tests or the urinalysis testing are not within the laboratory's reference ranges the volunteer can be included only on condition that the investigator judges that the deviations are not clinically significant.

Exclusion Criteria:

* History or suspicion of alcohol, barbiturate, amphetamine or narcotic abuse
* History of cardiac arrhythmias, bronchospastic or respiratory disease, cardiovascular, neurologic, renal, hepatic, endocrine, or immunologic disease
* Drug allergy to raclopride, paliperidone, or risperidone or any of its excipients
* Use of concomitant medication, except for paracetamol and hormonal contraceptives. All other medication must have been stopped at least 14 days before the first PET examination
* Received an experimental drug or used an experimental medical device within 30 days before the planned start of treatment
* Previously used an antipsychotic medication
* Previously participated in a PET study or measurement
* Had a significant loss of blood <1 month before the first PET examination
* Pregnant as confirmed by a positive beta-HCG test at screening and before the first PET examination, or breastfeeding
* Claustrophobia.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2003-03; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
to evaluate D2 receptor occupancy and plasma concentration of paliperidone at defined times after intake of a single dose of OROS paliperidone 6 mg

SECONDARY OUTCOMES:
to derive pharmacokinetic/pharmacodynamic relationships and the occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of dopamine type 2 (D2) receptor occupancy following a single oral dose of OROS paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=574&filename=CR004267_CSR.pdf